CLINICAL TRIAL: NCT05897580
Title: Impact of Community-Based Biofeedback Program on Drug Use and Mental Health Among People Experiencing Homelessness
Acronym: HRV-BF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Adeline Nyamathi, Distinguished Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20216820
Record Dates: First submitted 2023-05-12; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Heart Rate Variability
Keywords: heart rate variability; mental health; anxiety; depression; PTSD
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic | interventions — Health Promotion

STUDY DESIGN:
Intervention Model Description: Heart rate variability-biofeedback (HRV-BF) has been shown to decrease symptoms of stress, anxiety, depression, and PTSD, however HRV-BF has not been tested with the most vulnerable of populations, homeless adults
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart Rate Variability-Biofeedback (HRV-BF) (Experimental): Heart Rate Variability-Biofeedback (HRV-BF) is a process by which physiological markers such as heart rate, respiration, and HRV are measured and "fed" back to the person on a computer screen. Guided paced slowed breathing, a skill taught in HRV-BF, maximizes the natural acceleration of heart rate with inspiration and deceleration with expiration and produces a rhythmic stimulation of the vagus nerve, providing the basis for the overall increase in parasympathetic/vagal tone over time if practiced regularly.
  Interventions: Behavioral: Heart Rate Variability - Biofeedback (HRV-BF)
- Health Promotion (HP) (Active Comparator): The Health Promotion (HP) active control group was originally developed utilizing community-based participatory research elements, including the establishment of a Community Advisory Board (CAB), with community stakeholders, social service providers and academicians and a manualized program was developed for the HP program. The 8-week program focused on the most common physical chronic diseases PEH experience, and included discussions of hypertension, diabetes, heart disease and arthritis; total over eight weeks, along with full discussion and referrals provided based on needs expressed by PEH.
  Interventions: Behavioral: Health Promotion (HP)

INTERVENTIONS:
Behavioral: Heart Rate Variability - Biofeedback (HRV-BF) — The HRV-BF was delivered over 30 minutes once weekly for 8 weeks by our nurse-led Community Health Worker (RN/CHW) team trained to deliver scripted material created by a trained biofeedback practitioner on our study team. The weekly sessions included the use of a tablet device to share a 10-minute video which teaches the basic techniques and breathing practices of HRV-BF and guiding the participant through a 20-minute practice, using the techniques while watching their heart rate data in real time using an HRV-BF device, the EmWave Pro (HeartMath).
  Participants were also asked to complete daily practices on their own, without the HRV-BF device, for 10 minutes, twice a day, to reinforce topics and skills taught in videos. Practices logged by the participant were collected weekly by the CHW and referral to resources were provided.
  Arms: Heart Rate Variability-Biofeedback (HRV-BF)
Behavioral: Health Promotion (HP) — The HP active control group was delivered over 30 minutes, once weekly for 8 weeks by our nurse-led Community Health Worker team, trained to deliver scripted materialized content created. In the HP program, PEH were educated on common physical chronic diseases PEH experience, including hypertension, diabetes, heart disease and arthritis, along with referrals provided based on needs expressed by PEH.
  Arms: Health Promotion (HP)

SUMMARY:
The purpose of this randomized controlled trial was to compare the effectiveness of an HRV-BF intervention versus a health promotion active control intervention focused on improving mental health symptoms among people experiencing homelessness (PEH), who were residing in Skid Row, Los Angeles. In total, 40 PEH were randomized to either the HRV-BF or an active health promotion control group, and received 8 weekly, 30-minute sessions over a two month period, delivered by a nurse-led community health worker team. Dependent variables of HRV, mental health, anxiety, depression and PTSD were measured at baseline, the 8-week session, and/or 2-month follow up.

DETAILED DESCRIPTION:
In this pilot randomized controlled trial, conducted over one year, beginning in April 2021, 40 PEH were recruited from a larger sample of 100 PEH that were participating in a survey on COVID-19. Our outcomes were HRV and symptoms of anxiety, depression and PTSD.

Prior to the intervention, a Community Advisory Board (CAB) met to assess feasibility and acceptability of the HRV-BF program, which was presented in a theater-style approach. The CAB, composed of 6 PEH, and 3 healthcare providers, spoke quite favorably about the program, and provided exceptional feedback in terms of acceptability and feasibility in delivery logistics and cultural sensitivity. PEH shared the high levels of stress and anxiety they were experiencing; how helpful they perceived the program to be, the best timing for delivery, length of time for the intervention (under 60 minutes), and how to minimize attrition. Our study was approved by the Human Subjects Protection Committee at the University of California, Irvine and the University of California, Los Angeles.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* self-reported as residing in a homeless living condition during the previous night
* self-reported having used illicit substances or alcohol during the past year

Exclusion Criteria:

Persons who:

* exclusively spoke languages other than English or Spanish
* were unable to understand informed consent
* had cardiac deficiency, arrhythmias or pacemakers or who took medications affecting autonomic function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate Variability | Change Assessed during the resting 5-minute period at week 1 and week 8 sessions
  Commercially available, medical grade photodetector (photoplethysmography or PPG) sensor and accompanying HRV-BF software application (EmWave Pro Plus, HeartMath) will be used to collect interbeat interval data to produce standard measures of HRV including time-domain measures of SDNN (standard deviation of N-to-N intervals) and RMSSD (Root mean square of successive differences between normal heart beats). Both SDNN and RMSSD are measured in milliseconds (ms). RMSSD is most reflective of vagal tone and is our primary outcome measure.

SECONDARY OUTCOMES:
Mental Health Status | Baseline and 8 weeks
  Assessed by the Mental Health Inventory-5 (MHI-5) which has well-demonstrated reliability for detecting psychological disorders with reliabilities of .77 and .71 for women/men, respectively. Minimum = 5; Maximum = 30; Higher score means a better outcome.
Anxiety Symptoms | Baseline and 8 weeks
  Anxiety Symptoms were measured by the Generalized Anxiety Disorder -7, a self-report 7- item measure. Example items include "worrying too much about different things," and "trouble relaxing" (Endpoints 0=not at all; 3=nearly every day). Scores are summed. Severity of anxiety was determined with cut-off scores 5 (mild anxiety), 10 (moderate anxiety), and 15 (severe anxiety). Reliability α=0.87. Minimum = 0; Maximum = 21; Higher score means a worse outcome.
Depression Symptoms | Baseline and 8 weeks
  Depressive Symptoms were assessed by the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a brief, 9 question depression module from the full 26-item PHQ. Each of the 9 items address the Diagnostic and Statistical Manual of Mental Disorders (DSM) diagnostic criteria, rating them from "0" (not at all) to "3" (nearly every day). PHQ-9 not only makes criteria-based diagnoses of depressive disorders, but as well can determine severity, with scoring cut-offs for minimal (1-4), mild (5-9), moderate (10-14), moderately severe (15-19) and severe (20-27) depression. Reliability of the PHQ-9 is α=0.89. Minimum = 0; Maximum = 27; Higher score means a worse outcome.
Post Traumatic Stress Disorder (PTSD) | Baseline and 8 weeks
  PTSD was measured by means of the Post Traumatic Stress Disorder Checklist-5 (PCL-C), a 17-item screener for PTSD with cut points for symptomatic vs non-symptomatic; scores correlate highly with the Clinician Administered PTSD scale, r = .93.70 The PCL-C has high levels of validity,71 test-retest reliability (r = .96), and high internal consistency (α = .97). The self-report rating scale is 0-4 for each symptom: "Not at All" to "Extremely" (0-80). 5-point change is a minimum threshold for determining a treatment response, while a 10-point change is a minimum threshold for determining a clinically meaningful treatment response. Minimum = 17; Maximum = 85; Higher score means a worse outcome.
Drug and Alcohol Use | Baseline and 8 weeks
  Drug and Alcohol Use was assessed by the Texas Christian University (TCU) Drug History Form. It records the frequency of use of 16 drugs used over 12 months, such as heroin and other opiates, street methadone, cocaine, crack, methamphetamine, etc. Yes/No to each drug was assessed for use vs dependency. The total score ranges from 0 - 9; higher scores (> 3) correspond to the DSM 4 drug dependence diagnosis. Minimum = 0; Maximum = 11; Higher score means a worse outcome.
Physical Disease | Baseline and 8 weeks
  Physical Diseases was assessed by the self-reported comorbidity index (SCQ) for medical problem, treatment, and limitations. PEH were asked to respond if they have chronic health conditions (e.g., heart disease, high blood pressure, diabetes, osteoarthritis). Responses include "yes or no". In a previous PEH sample (N=150), Cronbach's α = .91.
  Physical Diseases was assessed by the self-reported comorbidity index (SCQ) for medical problem, treatment, and limitations. PEH were asked to respond if they have chronic health conditions (e.g., heart disease, high blood pressure, diabetes, osteoarthritis. Responses include "yes or no". In a previous PEH sample (N=150), Cronbach's α = .91. Minimum = 0; Maximum = 36; Higher score means a worse outcome.
Assessing Evidence of Drug Use in Urine | Baseline and 8 weeks
  Urinalysis: In addition, we conducted a urine assay which measures cannabis, methamphetamine, cocaine, and amphetamines. A five-panel Food and Drug Administration-approved urine test cup was used at baseline and 8 week follow-up. The test cup screened for metabolites of Amphetamines (1000 ng/mL), Cocaine (300 ng/mL), Methamphetamines (500 ng/mL), Opiates (2000 ng/mL), and Cannabis (THC) (50 ng/mL).

OTHER OUTCOMES:
Social Support | Baseline and 8 weeks
  Social support was measured by the Medical Outcome Study (MOS) Social Support Survey. The MOS is a 19-item instrument and includes four subscales: emotional and informational support; tangible support; positive social interaction; and affectionate support. The MOS uses a Likert-scale, with endpoints 1 (none of the time) to 5 (all of the time) that assesses availability of social support, with higher scores indicating more social support. An overall support index was also calculated.• Minimum = 0; Maximum = 100; Higher score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Amity Foundation, Los Angeles, Los Angeles, California
  - Downtown Women Center, Los Angeles, Los Angeles, California
  - Los Angeles Christian Health Centers (LACHC), Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berwick DM, Murphy JM, Goldman PA, Ware JE Jr, Barsky AJ, Weinstein MC. Performance of a five-item mental health screening test. Med Care. 1991 Feb;29(2):169-76. doi: 10.1097/00005650-199102000-00008. PMID 1994148
- [Background] Blackburn L, Owens GP. The effect of self efficacy and meaning in life on posttraumatic stress disorder and depression severity among veterans. J Clin Psychol. 2015 Mar;71(3):219-28. doi: 10.1002/jclp.22133. Epub 2014 Sep 30. PMID 25270887
- [Background] Forbes D, Creamer M, Biddle D. The validity of the PTSD checklist as a measure of symptomatic change in combat-related PTSD. Behav Res Ther. 2001 Aug;39(8):977-86. doi: 10.1016/s0005-7967(00)00084-x. PMID 11480838
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Laborde S, Mosley E, Thayer JF. Heart Rate Variability and Cardiac Vagal Tone in Psychophysiological Research - Recommendations for Experiment Planning, Data Analysis, and Data Reporting. Front Psychol. 2017 Feb 20;8:213. doi: 10.3389/fpsyg.2017.00213. eCollection 2017. PMID 28265249
- [Background] Leake B, Nyamathi A, Gelberg L. Reliability, validity, and composition of a subset of the Centers for Disease Control and Prevention acquired immunodeficiency syndrome knowledge questionnaire in a sample of homeless and impoverished adults. Med Care. 1997 Aug;35(8):747-55. doi: 10.1097/00005650-199708000-00001. PMID 9268248
- [Background] Lehrer P, Kaur K, Sharma A, Shah K, Huseby R, Bhavsar J, Sgobba P, Zhang Y. Heart Rate Variability Biofeedback Improves Emotional and Physical Health and Performance: A Systematic Review and Meta Analysis. Appl Psychophysiol Biofeedback. 2020 Sep;45(3):109-129. doi: 10.1007/s10484-020-09466-z. PMID 32385728
- [Background] McDonald SD, Calhoun PS. The diagnostic accuracy of the PTSD checklist: a critical review. Clin Psychol Rev. 2010 Dec;30(8):976-87. doi: 10.1016/j.cpr.2010.06.012. Epub 2010 Jul 6. PMID 20705376
- [Background] Nyamathi A. Comprehensive health seeking and coping paradigm. J Adv Nurs. 1989 Apr;14(4):281-90. doi: 10.1111/j.1365-2648.1989.tb03415.x. PMID 2661620
- [Background] Porges SW. The polyvagal perspective. Biol Psychol. 2007 Feb;74(2):116-43. doi: 10.1016/j.biopsycho.2006.06.009. Epub 2006 Oct 16. PMID 17049418
- [Background] Salem BE, Ma-Pham J. Understanding Health Needs and Perspectives of Middle-Aged and Older Women Experiencing Homelessness. Public Health Nurs. 2015 Nov-Dec;32(6):634-44. doi: 10.1111/phn.12195. Epub 2015 Mar 31. PMID 25832775
- [Background] Samuelson KW, Bartel A, Valadez R, Jordan JT. PTSD symptoms and perception of cognitive problems: The roles of posttraumatic cognitions and trauma coping self-efficacy. Psychol Trauma. 2017 Sep;9(5):537-544. doi: 10.1037/tra0000210. Epub 2016 Oct 13. PMID 27736138
- [Background] Sangha O, Stucki G, Liang MH, Fossel AH, Katz JN. The Self-Administered Comorbidity Questionnaire: a new method to assess comorbidity for clinical and health services research. Arthritis Rheum. 2003 Apr 15;49(2):156-63. doi: 10.1002/art.10993. PMID 12687505
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Wilkins KC, Lang AJ, Norman SB. Synthesis of the psychometric properties of the PTSD checklist (PCL) military, civilian, and specific versions. Depress Anxiety. 2011 Jul;28(7):596-606. doi: 10.1002/da.20837. Epub 2011 Jun 16. PMID 21681864
- [Background] Wingood GM, DiClemente RJ. The ADAPT-ITT model: a novel method of adapting evidence-based HIV Interventions. J Acquir Immune Defic Syndr. 2008 Mar 1;47 Suppl 1:S40-6. doi: 10.1097/QAI.0b013e3181605df1. PMID 18301133